CLINICAL TRIAL: NCT03030872
Title: Clinical Evaluation of CARESTREAM Vue PACS v12.2 MR Perfusion and Diffusion
Status: Completed | Type: Observational
Sponsor: Carestream Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AD0542
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-03

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Predicate software: Olea Sphere PACS with Perfusion and DWI Modules
- Investigational software: Vue PACS v12.2 Magnetic Resonance (MR) Perfusion and Diffusion Weighted Imaging
  Interventions: Device: Investigational software

INTERVENTIONS:
Device: Investigational software — The study evaluated retrospective de-identified cases that were processed after the imaging procedure had been completed (off-line) using a dedicated workstation.
  Groups: Investigational software

SUMMARY:
The objective of this study is to compare the diagnostic value of MR DSC-Perfusion (Perfusion Module), MR DWI (Diffusion Module) and MR DTI (Diffusion Module) in CARESTREAM Vue PACS ("investigational device") to the Olea Sphere PACS with Perfusion and DWI Modules ("predicate device"). Therefore, there will be several separate objectives depending on the type of acquisition:

DETAILED DESCRIPTION:
Carestream Health, Inc. will investigate the imaging performance of the CARESTREAM Vue PACS v12.2 Magnetic Resonance (MR) Perfusion and Diffusion Weighted Imaging ("investigational device") performance. Evaluation of MR Dynamic Susceptibility Contrast-Enhanced Perfusion Weighted Imaging (DSC-Perfusion), MR Diffusion Weighted Imaging (DWI) and MR Diffusion Tensor Imaging (DTI) was compared to the predicate device, the Olea Sphere PACS with Perfusion and DWI Modules. MR DSC-Perfusion of the brain is a method for evaluating blood flow in the brain and producing optimized parametric maps that help visualize this blood flow. MR DWI is a method to evaluate the motion of water molecules within bodily tissues. MR DTI is an extension of DWI that allows extraction of the diffusion tensor. The purpose of this study is to demonstrate equivalent clinical quality between the investigational and predicate devices using a radiologist evaluation of key metrics which are applicable to MR DSC-Perfusion, MR DWI, and MR DTI images.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective patient MR DSC-Perfusion cases with subject/patient 18 years of age or older.
* Retrospective patient MR DWI with subject/patient 18 years of age or older.
* Retrospective patient MR DTI cases with subject/patient 18 years of age or older.
* Informed consent is not required if waiver of consent is approved by the hospital IRB/Ethics Committee

Exclusion Criteria:

* Low quality images, or images that are not clinically acceptable for clinical diagnostic reading as determined by the Principal Investigator
* Subject less than 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of retrospective de-identified adult patient MR DSC-Perfusion, DWI, and DTI (if available) cases collected under Ethics Committee/IRB approval. The Ethics Committee/IRB submission will request a waiver of patient informed consent in compliance with local country regulations, and must meet the study inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-01-07 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic value comparison of Carestream Vue PACS v12.2 MR Perfusion and Diffusion (investigational software) images to the Olea Shere PACS with Perfusion and DWI Modules (predicate software) images. | January 2017
  Diagnostic value of investigational images compared to the diagnostic value of predicate images as assessed by a radiologist evaluation of key metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Pate, MS, RN, Study Director — Senior Manager Clinical Affairs

IPD SHARING:
Plan to Share IPD: No